CLINICAL TRIAL: NCT02418858
Title: Randomized Controlled Clinical Trial Comparing Functional Outcomes of Awake vs. Asleep Deep Brain Stimulation (DBS) for Essential Tremor
Brief Title: Functional Outcomes of Awake vs. Asleep Deep Brain Stimulation (DBS) for Essential Tremor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subject enrollment
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 14BN146
Record Dates: First submitted 2015-03-24; First posted 2015-04-16 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Essential Tremor
Keywords: Essential tremor; DBS
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Awake DBS Surgery (Active Comparator): Deep brain stimulation surgery: Essential tremor patients undergoing traditional "awake" DBS surgery utilizing microelectrode recordings and intraoperative stimulation.
  Interventions: Procedure: Deep Brain Stimulation surgery
- Asleep DBS Surgery (Active Comparator): Deep brain stimulation surgery: Essential tremor patients undergoing DBS surgery under general anesthesia utilizing intraoperative imaging to verify the stereotactic accuracy of DBS electrode placement at the time of surgery.
  Interventions: Procedure: Deep Brain Stimulation surgery

INTERVENTIONS:
Procedure: Deep Brain Stimulation surgery — Deep Brain Stimulation surgery awake vs. asleep
  Other Names: DBS

SUMMARY:
Recently, there has been increasing interest in performing DBS under general anesthesia, where the stimulated targets are located anatomically (i.e. on MRI) rather than physiologically via microelectrode recordings and intra-operative test stimulation. This technology has been termed "asleep" DBS and is performed with the patient under general anesthesia. Intraoperative imaging is utilized to verify the stereotactic accuracy of DBS electrodes placement at the time of surgery. Because stereotactic accuracy (and surgical safety) is the surgical endpoint, there is no need for the patient to be awake during the procedure.

DETAILED DESCRIPTION:
Traditional DBS is performed without general anesthesia with the patient awake. Local anesthetic is used to numb the skin and tissue where the incision is made, and the patients are given mild sedatives to alleviate anxiety and discomfort. Essential tremor (ET) patients undergo intra-operative test stimulation to refine the lead location and ensure the absence of sustained side effects. This can result in multiple brain penetrations during lead placement, and the entire procedure may last anywhere from 4-6 hours on average. The concept of being awake during brain surgery provokes significant anxiety and fear in some patients.

Recently, there has been increasing interest in performing DBS under general anesthesia, where the stimulated targets are located anatomically (i.e. on MRI) rather than physiologically via microelectrode recordings and intra-operative test stimulation. This technology has been termed "asleep" DBS and is performed with the patient under general anesthesia. Intraoperative imaging is utilized to verify the stereotactic accuracy of DBS electrodes placement at the time of surgery. Because stereotactic accuracy (and surgical safety) is the surgical endpoint, there is no need for the patient to be awake during the procedure.

If asleep DBS produces clinical results equivalent to awake DBS surgery, the possible advantages include shorter surgical time, improved patient comfort, better access to DBS for patients, and cost savings for the hospital.

To date (August 2011 - September 2014), 157 patients have undergone asleep DBS surgery and 141 patients have undergone traditional awake DBS surgery. ET patients constitute 76 of the total surgeries - 50 patients underwent awake surgery and 26 underwent asleep surgery. The safety and efficacy of the two approaches to DBS surgery have been equivalent, and we are at a position of equipoise with regard to what to offer to patients. To date, there have been no randomized, controlled clinical trials comparing the efficacy and functional outcomes of the two DBS methods for patients with the diagnosis of Essential tremor. The purpose of the proposed study is to demonstrate that the functional outcomes of the "asleep" technique are not inferior to those reported for traditional "awake" DBS technique. The primary data points for this study will include three month functional outcomes using accepted outcome metrics for ET, including an objective tremor rating scale (Fahn-Tolosa-Marin Tremor Rating Scale), a tremor Activities of Daily Living (ADL) questionnaire (Bain and Findley Tremor ADL scale), and a tremor quality of life questionnaire : Quality of Life in Essential Tremor Questionnaire [QUEST]). Parkinson Meter and Life Pulse tremor readings (two iPhone accelerometer applications) will also be collected. . Patients who elect to participate in this trial will undergo a routine pre-operative neurocognitive evaluation consisting of the following routine evaluative tests: Wechsler Test of Adult Reading, Mattis Dementia Rating Scale 2nd Edition, Wechsler Abbreviate Scale of Intelligence 2nd Edition; Wechsler Memory Scale 3rd edition, Digit Span, Stroop Neuropsychological Screening Test, Trail Making Test, Wisconsin Card Sorting Test, Controlled Oral Word Association Test, Animal Naming, Boston Naming Test, Wechsler Memory Scale 4th Edition, Logical Memory, Hopkins Verbal Learning Test - Revised, Brief Visuospatial Memory Test - Revised, Hooper visual Organization Test, Judgment of Line Orientation, Beck Depression Inventory, Beck Anxiety Inventory, Epworth Sleepiness Scale. The subjects will then be randomized to 2 groups by using random numbers in an envelope system. We anticipate that 120 total patients will need to be enrolled in this pilot study (60 awake, 60 asleep), and thus the numbers 1-120 will be placed in envelopes. An odd number will correspond to the awake DBS procedure, and an even number will indicate an asleep DBS procedure. The null hypothesis is that asleep DBS results in inferior tremor ratings 3-months after surgery when compared to awake DBS. Our secondary aim will be to evaluate any cognitive changes associated with DBS surgery selection (awake vs. asleep) in ET patients. Current standard of care for patient selection in DBS focuses primarily on the evaluation of motor symptoms and currently there is no guidance for how a patients' DBS surgery selection (awake vs. asleep) would impact on subsequent neurocognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Essential Tremor diagnosed by criteria listed in the Consensus statement of the Movement Disorders Society on Tremor
* Age 18 - 85 years of age
* Motor skills allowing for capability to complete evaluations
* Medically cleared for undergoing anesthesia and DBS surgery

Exclusion Criteria:

* Dementia per DSM-V criteria
* Medical or other condition precluding MRI
* History of supraspinal CNS disease other than Essential Tremor
* Alcohol use of more than 4 drinks per day
* Pregnancy
* History of suicide attempt
* Currently uncontrolled clinically significant depression (BDI>20)
* History of schizophrenia, delusions, or currently uncontrolled visual hallucinations

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Functional Outcomes | 12 weeks post-operatively
  The primary data points for this study will include three month functional outcomes using accepted outcome metrics for ET, including an objective tremor rating scale (Fahn-Tolosa-Marin Tremor Rating Scale), a tremor ADL questionnaire (Bain and Findley Tremor ADL scale) for comparison to preoperative scores.
Quality of Life Assessment | 12 week post-operatively
  Quality of life in Essential Tremor [QUEST] questionnaire will be collected again for comparison to preoperative scores.

SECONDARY OUTCOMES:
Neurocognitive Function | 6 months post-operatively
  Neurocognitive evaluation consisting of the following routine evaluative tests: Wechsler Test of Adult Reading, Mattis Dementia Rating Scale 2nd Edition, Wechsler Abbreviate Scale of Intelligence 2nd Edition; Wechsler Memory Scale 3rd edition, Digit Span, Stroop Neuropsychological Screening Test, Trail Making Test, Wisconsin Card Sorting Test, Controlled Oral Word Association Test, Animal Naming, Boston Naming Test, Wechsler Memory Scale 4th Edition, Logical Memory, Hopkins Verbal Learning Test - Revised, Brief Visuospatial Memory Test - Revised, Hooper visual Organization Test, Judgment of Line Orientation, Beck Depression Inventory, Beck Anxiety Inventory, Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease, Apathy Evaluation Scale; Epworth Sleepiness Scale.

OTHER OUTCOMES:
Tremor Reduction | 12 weeks post-operatively
  Parkinson Meter and Life Pulse tremor readings will be collected for comparison to preoperative scores.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Ponce, MD, Principal Investigator — Barrow Neurological Institute / St. Joseph's Hospital and Medical Center
Locations (1):
- Barrow Neurological Institute / St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Background] Bain PG, Findley LJ, Atchison P, Behari M, Vidailhet M, Gresty M, Rothwell JC, Thompson PD, Marsden CD. Assessing tremor severity. J Neurol Neurosurg Psychiatry. 1993 Aug;56(8):868-73. doi: 10.1136/jnnp.56.8.868. PMID 8350102
- [Background] Elble R, Bain P, Forjaz MJ, Haubenberger D, Testa C, Goetz CG, Leentjens AF, Martinez-Martin P, Pavy-Le Traon A, Post B, Sampaio C, Stebbins GT, Weintraub D, Schrag A. Task force report: scales for screening and evaluating tremor: critique and recommendations. Mov Disord. 2013 Nov;28(13):1793-800. doi: 10.1002/mds.25648. Epub 2013 Sep 3. PMID 24038576
- [Background] Flora ED, Perera CL, Cameron AL, Maddern GJ. Deep brain stimulation for essential tremor: a systematic review. Mov Disord. 2010 Aug 15;25(11):1550-9. doi: 10.1002/mds.23195. PMID 20623768
- [Background] Troster AI, Pahwa R, Fields JA, Tanner CM, Lyons KE. Quality of life in Essential Tremor Questionnaire (QUEST): development and initial validation. Parkinsonism Relat Disord. 2005 Sep;11(6):367-73. doi: 10.1016/j.parkreldis.2005.05.009. PMID 16103000
- [Background] Ostrem JL, Galifianakis NB, Markun LC, Grace JK, Martin AJ, Starr PA, Larson PS. Clinical outcomes of PD patients having bilateral STN DBS using high-field interventional MR-imaging for lead placement. Clin Neurol Neurosurg. 2013 Jun;115(6):708-12. doi: 10.1016/j.clineuro.2012.08.019. Epub 2012 Sep 1. PMID 22944465
- [Background] Burchiel KJ, McCartney S, Lee A, Raslan AM. Accuracy of deep brain stimulation electrode placement using intraoperative computed tomography without microelectrode recording. J Neurosurg. 2013 Aug;119(2):301-6. doi: 10.3171/2013.4.JNS122324. Epub 2013 May 31. PMID 23724986
- [Background] Weaver FM, Follett K, Stern M, Hur K, Harris C, Marks WJ Jr, Rothlind J, Sagher O, Reda D, Moy CS, Pahwa R, Burchiel K, Hogarth P, Lai EC, Duda JE, Holloway K, Samii A, Horn S, Bronstein J, Stoner G, Heemskerk J, Huang GD; CSP 468 Study Group. Bilateral deep brain stimulation vs best medical therapy for patients with advanced Parkinson disease: a randomized controlled trial. JAMA. 2009 Jan 7;301(1):63-73. doi: 10.1001/jama.2008.929. PMID 19126811
- [Background] Pezeshkian P, DeSalles AA, Gorgulho A, Behnke E, McArthur D, Bari A. Accuracy of frame-based stereotactic magnetic resonance imaging vs frame-based stereotactic head computed tomography fused with recent magnetic resonance imaging for postimplantation deep brain stimulator lead localization. Neurosurgery. 2011 Dec;69(6):1299-306. doi: 10.1227/NEU.0b013e31822b7069. PMID 21725253
- [Background] Alexander E 3rd, Kooy HM, van Herk M, Schwartz M, Barnes PD, Tarbell N, Mulkern RV, Holupka EJ, Loeffler JS. Magnetic resonance image-directed stereotactic neurosurgery: use of image fusion with computerized tomography to enhance spatial accuracy. J Neurosurg. 1995 Aug;83(2):271-6. doi: 10.3171/jns.1995.83.2.0271. PMID 7616273
- [Background] Papanastassiou V, Rowe J, Scott R, Silburn P, Davies L, Aziz T. Use of the Radionics Image Fusiontrade mark and Stereoplantrade mark programs for target localization in functional neurosurgery. J Clin Neurosci. 1998 Jan;5(1):28-32. doi: 10.1016/s0967-5868(98)90197-7. PMID 18644283
- [Background] Kooy HM, van Herk M, Barnes PD, Alexander E 3rd, Dunbar SF, Tarbell NJ, Mulkern RV, Holupka EJ, Loeffler JS. Image fusion for stereotactic radiotherapy and radiosurgery treatment planning. Int J Radiat Oncol Biol Phys. 1994 Mar 30;28(5):1229-34. doi: 10.1016/0360-3016(94)90499-5. PMID 8175410